CLINICAL TRIAL: NCT01554462
Title: The Effects of Eicosapentaenoic Acid (EPA)/ Docosahexaenoic Acid (DHA) Supplementation on Cognitive Control in Children With Attention Deficit Hyperactivity Disorder (ADHD)
Brief Title: The Effects of EPA/DHA Supplementation on Cognitive Control in Children With ADHD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Unilever R&D (Industry)
Collaborators: UMC Utrecht (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: 08033V
Record Dates: First submitted 2012-02-28; First posted 2012-03-15 (Estimated); Last update posted 2013-12-11 (Estimated); Status verified 2013-12

CONDITIONS: Attention Deficit Hyperactivity Disorder; Healthy
Keywords: Attention; Cognitive control; ADHD; Healthy; EPA; Eicosapentaenoic acid; DHA; Docosahexaenoic acid; PUFA; Omega-3
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity | interventions — Eicosapentaenoic Acid; Docosahexaenoic Acids; Fatty Acids, Monounsaturated

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- ADHD active (Active Comparator): 4 month intervention with EPA/DHA in ADHD group
  Interventions: Dietary Supplement: Eicosapentaenoic acid / Docosahexaenoic acid
- ADHD Placebo (Placebo Comparator): 4 month dietary intervention with placebo in ADHD group
  Interventions: Dietary Supplement: Placebo dietary intervention (MUFA) in ADHD group
- Active Healthy control (Active Comparator): 4 month dietary intervention with DHA/EPA in healthy control group
  Interventions: Dietary Supplement: Eicosapentaenoic acid / Docosahexaenoic acid
- Healthy placebo (Placebo Comparator): 4 month dietary intervention with placebo in healthy control group
  Interventions: Dietary Supplement: Placebo dietary intervention (MUFA) in healthy control group

INTERVENTIONS:
Dietary Supplement: Eicosapentaenoic acid / Docosahexaenoic acid — 650 mg EPA + 650 mg DHA daily
  Other Names: EPA; DHA
  Arms: ADHD active
Dietary Supplement: Placebo dietary intervention (MUFA) in ADHD group — Placebo contains mono-unsaturated fatty acids (MUFA) in stead of poly-unsaturated fatty acids (PUFA), same energy value
  Other Names: Mono Unsaturated Fatty Acid; Poly Unsaturated Fatty Acid
  Arms: ADHD Placebo
Dietary Supplement: Eicosapentaenoic acid / Docosahexaenoic acid — 650 mg EPA and 650 mg DHA daily
  Other Names: EPA; DHA
  Arms: Active Healthy control
Dietary Supplement: Placebo dietary intervention (MUFA) in healthy control group — Placebo contains MUFA in stead of PUFA, same energy value
  Other Names: Mono Unsaturated Fatty Acids
  Arms: Healthy placebo

SUMMARY:
Forty children with and 40 children without Attention deficit Hyperactivity Disorder (ADHD) receive Docosahexaenoic Acid (DHA) and Eicosapentaenoic Acid (EPA) or placebo via a dietary intervention. Cognitive control functions are measured with functional Magnetic Resonance Imaging (MRI) before and after the intervention. Behavioural change is monitored with behavioural scales.

ELIGIBILITY:
Inclusion Criteria:

Inclusion criteria for subjects with ADHD

1. 8-12 year old boys
2. Diagnostic and Statistical Manual 4th edition (DSM-IV (APA, 1994)) diagnosis of ADHD, according to Diagnostic Interview Schedule for Children (DISC)
3. Scores in the clinical range on the Child Behaviour Checklist (CBCL) and Teacher Rating Form(TRF)
4. Ability to speak and comprehend Dutch.
5. Used to daily consumption of margarine

Inclusion criteria for controls

1. 8-12 year old boys
2. No DSM-IV (APA, 1994) diagnosis, according to DISC interview
3. No scores in the clinical range on the Child Behaviour Checklist (CBCL) and Teacher Rating Form (TRF)
4. Ability to speak and comprehend Dutch. 5 Used to daily consumption of margarine

Exclusion Criteria:

1. mental retardation (IQ < 70)
2. major illness of the cardiovascular, the endocrine, the pulmonary or the gastrointestinal system
3. presence of metal objects in or around the body (pacemaker, dental braces)
4. history of or present neurological disorder
5. regular use of n-3 or n-6 fatty acid dietary supplements, products fortified with EPA or DHA, a regular diet high in fatty fish (= 1 serving per week) or participation in intervention studies or (school-) health programs in the four months prior to study participation.

Ages: 8 Years to 12 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 79 (Actual)
Dates: Start 2009-01; Primary Completion 2013-01 (Actual); Study Completion 2013-01 (Actual)

PRIMARY OUTCOMES:
Cognitive control task - functional MRI | change over 16 week intervention period (pre/post)

SECONDARY OUTCOMES:
Behavioural scales: - Child Behaviour Checklist (CBCL) / Teacher Report Form (TRF) - Strengths and Weaknesses of ADHD-symptoms and Normal behaviour (SWAN) questionnaire | Change over 16 week intervention period (pre/post)
Fatty acids status from cheek cells (swabs) | Change over 16 week intervention period (pre/post)

CONTACTS AND LOCATIONS:
Overall Officials: Marco Hoeksma, PhD, Study Director — Unilever Research Vlaardingen; Sarah Durston, PhD, Principal Investigator — UMC Utrecht
Locations (1):
- Utrecht University Medical Center; Child and adolescent psychiatry, Utrecht, Netherlands

REFERENCES:
- [Derived] Gillies D, Leach MJ, Perez Algorta G. Polyunsaturated fatty acids (PUFA) for attention deficit hyperactivity disorder (ADHD) in children and adolescents. Cochrane Database Syst Rev. 2023 Apr 14;4(4):CD007986. doi: 10.1002/14651858.CD007986.pub3. PMID 37058600
- [Derived] Bos DJ, Oranje B, Veerhoek ES, Van Diepen RM, Weusten JM, Demmelmair H, Koletzko B, de Sain-van der Velden MG, Eilander A, Hoeksma M, Durston S. Reduced Symptoms of Inattention after Dietary Omega-3 Fatty Acid Supplementation in Boys with and without Attention Deficit/Hyperactivity Disorder. Neuropsychopharmacology. 2015 Sep;40(10):2298-306. doi: 10.1038/npp.2015.73. Epub 2015 Mar 19. PMID 25790022